CLINICAL TRIAL: NCT03047564
Title: Metal Ion Concentration and Clinical Outcome Between Coated and Uncoated TKA
Brief Title: Metal Ion Concentration Between Coated and Uncoated TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Mathys Ltd Bettlach (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKAcoated
Record Dates: First submitted 2017-01-24; First posted 2017-02-09 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2021-02

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Arthroplasty; Total Knee Replacement; Outcome; Metal ion concentration; Results
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomization to one of two implants
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coated Total Knee Arthroplasty (Experimental): Implantation of a coated Total Knee Arthroplasty
  Interventions: Device: Coated Total Knee Arthroplasty
- Standard Total Knee Arthroplasty (Active Comparator): Implantation of a Standard Total Knee Arthroplasty
  Interventions: Device: Standard Total Knee Arthroplasty

INTERVENTIONS:
Device: Coated Total Knee Arthroplasty — Implantation of a coated Total Knee Arthroplasty
  Arms: Coated Total Knee Arthroplasty
Device: Standard Total Knee Arthroplasty — Implantation of a Standard Total Knee Arthroplasty
  Arms: Standard Total Knee Arthroplasty

SUMMARY:
Metal ion release from metal implants may have side effects. It can be reduced by coating of the implant. This study compares coated and uncoated TKA.

DETAILED DESCRIPTION:
Patients are randomized to receive a coated or uncoated TKA. Patients are assessed before surgery, after 3 month, 1 year and 5 years.

Blood samples are collected in 7.5 ml S-Monovette® tubes (for trace metal analysis, Sarstedt AG, Germany) using a specific steel needle for trace metal analysis (Sarstedt AG, Germany). Within one hour, plasma was separated by centrifugation at 2500g for ten minutes. Samples were stored at -20°C before being analysed for chromium, cobalt, molybdenum and nickel content using a graphite furnace atomic absorption spectrometer Z-8270 with Polarisation-Zeeman-Absorption (Hitachi Ltd., Japan). The accuracy and precision of the method is validated to < 10% using the control materials SeronormTM Trace Elements Serum (SERO AS, Norway). The detection limit of the method is estimated at 0.5µg/l for chromium, cobalt and molybdenum, 1.0µg/l for nickel (mean + 3 standard deviations from buffer). All probes having ion levels below the detection limit were adjusted to 0.25µg/l for chromium, cobalt and molybdenum and 0.5µg/l for nickel.

Clinical outcome is measured with the Knee Society Score, Oxford Knee Score, Short-Form 36 and University of Los Angeles Activity Score.

ELIGIBILITY:
Inclusion Criteria:

* indication to TKA
* no other metal implant

Exclusion Criteria:

* no informed consent
* not able to understand study and/or questionnaires
* Need of a higher constrained implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Metal Ions (Cobalt, Chromium, Molydenum, Nickel) | before surgery, 1 year, 5 years
  Change in Serum Metal Ion concentrations 1 and 5 years after surgery

SECONDARY OUTCOMES:
Function | before surgery, 3 month, 1 year, 5 years
  Knee Society Score
Patient Reported Outcome | before surgery, 3 month, 1 year, 5 years
  Oxford Knee Score
Health-related Quality of Life | before surgery, 3 month, 1 year, 5 years
  SF 36
Activity | before surgery, 3 month, 1 year, 5 years
  UCLA activity score

OTHER OUTCOMES:
Adverse Events | through study completion, in average 5 years
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Lützner, MD, Principal Investigator — University Hospital Carl Gustav Carus

IPD SHARING:
Plan to Share IPD: Undecided